CLINICAL TRIAL: NCT02875405
Title: The Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery
Acronym: PALACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1502015867
Record Dates: First submitted 2016-07-25; First posted 2016-08-23 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: postoperative; pericardiotomy; prevention; cardiac surgery; left; posterior
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received pericardiotomy (Experimental): Patient will receive a posterior left pericardiotomy at the time of surgery
  Interventions: Procedure: Posterior left pericardiotomy
- No Pericardiotomy (No Intervention): Patient will not receive posterior left pericardiotomy.

INTERVENTIONS:
Procedure: Posterior left pericardiotomy — Patient will receive a posterior left sided pericardiotomy. The incision will be made posterior to the phrenic nerve and run from the inferior left pulmonary vein to the diaphragm.
  Arms: Received pericardiotomy

SUMMARY:
The purpose of this study is to determine if preforming a posterior left pericardiotomy prevents atrial fibrillation after cardiac surgery.

DETAILED DESCRIPTION:
Post-operative atrial fibrillation (POAF) is a common complication of cardiac surgery which is observed in 30-40% of patients. POAF may cause stroke, systemic embolism or cardiac failure and Its detection mandates for additional treatment with variable combinations of drugs to control cardiac rate or rhythm, anticoagulation, and electrical cardioversion, with their side effects and complications. As a result, POAF prolongs hospital stay and increases the costs of hospitalization. Several strategies aimed at reducing the incidence of POAF have been investigated, including beta-blockers, amiodarone, and statins, with unsatisfactory results. Posterior left pericardiotomy has been associated with a reduction in the incidence of POAF in a few studies. However, these studies are flawed by methodological limitations in terms of sample size, inclusion/exclusion criteria, randomization procedure, and suboptimal electrocardiographic monitoring strategies. Moreover, posterior left pericardiotomy requires additional operative time and is associated with procedure-specific complications. As a result, current evidence on posterior pericardiectomy failed to translate into changes in clinical practice and the incidence of POAF remains high.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients admitted to the department of cardiothoracic surgery of the NYPH-WCMC will be screened for enrollment.

Exclusion Criteria:

* preoperative non-sinus rhythm
* history of previous atrial arrhythmia of any type
* reoperations
* mitral or tricuspid valve disease
* surgery of the descending thoracic or thoracoabdominal aorta
* need for hypothermic circulatory arrest
* off pump operation
* urgent/emergent presentation
* disease of the left pleura or previous left thoracotomy
* chest deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Postoperative Atrial Fibrillation (POAF) | During hospitalization, approximately 5 days
  POAF occurrences are defined as any irregular heart rhythm, without detectable P-wave, that lasts more than 30 seconds.

SECONDARY OUTCOMES:
Duration of Postoperative Atrial Fibrillation (POAF) | During hospitalization, approximately 5 days
  Time spent in atrial fibrillation (seconds), defined as the time from the first evidence of atrial fibrillation to the first evidence of sinus rhythm restoration on cardiac monitoring strips or standard electrocardiograms (EKG)
Duration of Hospitalization | During hospitalization, up to 100 days after surgery
  Time (hours) spent in hospital after surgery completion

CONTACTS AND LOCATIONS:
Overall Officials: Leonard N Girardi, MD, Principal Investigator — Weill Cornell Medical College New York Presbyterian Hospital; Mario F Gaudino, MD, Study Chair — Weill Cornell Medical College New York Presbyterian Hospital
Locations (1):
- Weil Cornell Medical College Department of Cardiothoracic Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biancari F, Mahar MA. Meta-analysis of randomized trials on the efficacy of posterior pericardiotomy in preventing atrial fibrillation after coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2010 May;139(5):1158-61. doi: 10.1016/j.jtcvs.2009.07.012. Epub 2009 Aug 18. PMID 19691996
- [Result] Kaleda VI, McCormack DJ, Shipolini AR. Does posterior pericardiotomy reduce the incidence of atrial fibrillation after coronary artery bypass grafting surgery? Interact Cardiovasc Thorac Surg. 2012 Apr;14(4):384-9. doi: 10.1093/icvts/ivr099. Epub 2012 Jan 9. PMID 22235005
- [Derived] Gaudino M, Harik L, Redfors B, Sandner S, Alexander JH, Di Franco A, Dimagli A, Weinsaft J, Perezgrovas-Olaria R, Soletti GJ, Lau C, Mack C, Girardi L. The Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery-Extended Follow-Up study (PALACS-EF): rationale and design. Eur Heart J Open. 2023 Nov 17;3(6):oead118. doi: 10.1093/ehjopen/oead118. eCollection 2023 Nov. PMID 38035038
- [Derived] Rong LQ, Di Franco A, Rahouma M, Dimagli A, Chan J, Lopes AJ, Kim J, Sanna T, Devereux RB, Delgado V, Weinsaft JW, Crea F, Alexander JH, Gillinov M, DiMaio JM, Pryor KO, Girardi L, Gaudino M. Postoperative pericardial effusion, pericardiotomy, and atrial fibrillation: An explanatory analysis of the PALACS trial. Am Heart J. 2023 Jun;260:113-123. doi: 10.1016/j.ahj.2023.03.001. Epub 2023 Mar 18. PMID 36934978
- [Derived] Gaudino M, Sanna T, Ballman KV, Robinson NB, Hameed I, Audisio K, Rahouma M, Di Franco A, Soletti GJ, Lau C, Rong LQ, Massetti M, Gillinov M, Ad N, Voisine P, DiMaio JM, Chikwe J, Fremes SE, Crea F, Puskas JD, Girardi L; PALACS Investigators. Posterior left pericardiotomy for the prevention of atrial fibrillation after cardiac surgery: an adaptive, single-centre, single-blind, randomised, controlled trial. Lancet. 2021 Dec 4;398(10316):2075-2083. doi: 10.1016/S0140-6736(21)02490-9. Epub 2021 Nov 14. PMID 34788640
- [Derived] Abouarab AA, Leonard JR, Ohmes LB, Lau C, Rong LQ, Ivascu NS, Pryor KO, Munjal M, Crea F, Massetti M, Sanna T, Girardi LN, Gaudino M. Posterior Left pericardiotomy for the prevention of postoperative Atrial fibrillation after Cardiac Surgery (PALACS): study protocol for a randomized controlled trial. Trials. 2017 Dec 13;18(1):593. doi: 10.1186/s13063-017-2334-4. PMID 29237510